CLINICAL TRIAL: NCT02588768
Title: Phototherapy (With a Combination of Super-pulsed Laser and LEDs) in a Field Test With High-level Rugby Players
Brief Title: Photobiomodulation Therapy in a Field Test With High-level Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Multi Radiance Medical (Industry); São José Rugby Club (Other)
Responsible Party: Principal Investigator, Adriane Aver Vanin, PhD candidate, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CEP-665.347
Record Dates: First submitted 2015-10-24; First posted 2015-10-28 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: High-level Rugby Athletes; Performance; Recovery
Keywords: Low-level laser therapy; Light emitting diodes; Rugby; Field test; Photobiomodulation
MeSH Terms: interventions — Low-Level Light Therapy; Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active PBMT (Active Comparator): Active PBMT was applied employing MR4 Laser Therapy Systems outfitted with LaserShower 50 4D emitters (both manufactured by Multi Radiance Medical, Solon - OH, USA). The cluster style emitter contains 12 diodes comprising of four super-pulsed laser diodes (905 nm, 0.3125 mW average power, and 12.5 W peak power for each diode), four red LED diodes (640 nm, 15 mW average power for each diode), and four infrared LEDs diodes (875 nm, 17.5 mW average power for each diode).
  Interventions: Device: Photobiomodulation therapy (Phototherapy)
- Placebo PBMT (Placebo Comparator): Placebo PBMT was applied using the same device that emitted the same sounds and light, but with no effective irradiation.
  Interventions: Device: Photobiomodulation therapy (Phototherapy)

INTERVENTIONS:
Device: Photobiomodulation therapy (Phototherapy) — PBMT was applied employing MR4 Laser Therapy Systems manufactured by Multi Radiance Medical, Solon - OH, USA. The cluster emitter contains 12 diodes with four super-pulsed laser diodes (905 nm, 0.3125 mW average power, and 12.5 W peak power for each diode), four red LED diodes (640 nm, 15 mW average power for each diode), and four infrared LEDs diodes (875 nm, 17.5 mW average power for each diode). It was applied in direct contact with the skin to 9 sites on extensor muscles of the knee, 6 sites on knee flexors of the knee, and 2 sites on the calf of both lower limbs. To ensure blinding, the device emitted the same sounds and regardless of the programmed mode (active or placebo).
  Other Names: Photobiomodulation therapy (PBMT)

SUMMARY:
Background/Aim: While growing evidence supports the use of photobiomodulation therapy (PBMT) for performance and recovery enhancement, there have only been laboratory-controlled studies. Therefore, the aim of this study was to analyze the effects of PBMT in performance and recovery of high-level rugby players during an anaerobic field test.

Methods: It is a randomized, crossover, double-blinded, placebo-controlled trial. Twelve male high-level rugby athletes were recruited in this study. No intervention was performed before the Bangsbo Sprint Test (BST) at familiarization phase (week 1). At weeks 2 and 3, pre-exercise PBMT or placebo were randomly applied to each athlete. PBMT/placebo irradiation was performed at 17 sites of each lower limb, employing a cluster with 12 diodes (4 laser diodes of 905nm, 4 LED diodes of 875nm, and 4 LED diodes of 640nm, 30J per site - manufactured by Multi Radiance Medical™). Average time of sprints, best time of sprints, and fatigue index were obtained from BST. Blood lactate levels were assessed at baseline, and at 3, 10, 30 and 60 minutes after BST. Athletes' perceived fatigue was also assessed through a questionnaire.

DETAILED DESCRIPTION:
All exercise tests were conducted in an enclosed soccer/rugby field. The three test phases, administered one week apart, were performed on the same day of the week (Tuesday) and time (1-5pm). The average temperature inside the building during the trials ranged from 26°C to 28°C. At first stage (exercise test 1) all athletes performed the Bangsbo Sprint Test (BST) to familiarization with the procedure. No interventions or comparators were applied before this test. However, at the second and third stages (exercise tests 2 and 3, respectively) either a placebo or active PBMT was applied according to randomization. Blood samples were collected from the athlete's fingertips prior to stretching and warming-up (baseline), and at 3, 10, 30 and 60 minutes after BST at each of the three study stages/phase (exercise tests). After blood sample collection (to establish baseline), a warm-up comprised of low-intensity activities such as dynamic stretches and low-intensity short running were performed by each athlete. Following the warm-up and cool down period, either the active or placebo comparator was applied to the athlete according to the randomization procedure for the second test. For the third test, the other comparator was utilized to complete the cross over design. A quick perception of fatigue survey was administered following each test.

ELIGIBILITY:
Inclusion Criteria:

* high-level athletes from São José Rugby Club (Brazil)

Exclusion Criteria:

* Athlete would be excluded if the participant presented any skeletal muscle injury
* if athlete took any nutritional supplement or pharmacological agent
* if the athlete presented signs and symptoms of any disease (i.e., neurological, inflammatory, pulmonary, metabolic, oncologic), and
* if the athlete had history of cardiac arrest that could limit performance of high-intensity exercises

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Bangsbo Sprint Test (BST) - Average Time (sec) | The test was performed for three weeks, once a week, on the same day and time of the week.
  The Average Time of sprints performed during entire test (ST mean). This is the one of the variables from BST to evaluate performance.
Bangsbo Sprint Test (BST) - Best Time (sec) | The test was performed for three weeks, once a week, on the same day and time of the week.
  The fastest (best) time (ST best) among the seven sprints performed at each test. One of the variables from BST to evaluate performance.
Bangsbo Sprint Test (BST) - Fatigue Index (%) | The test was performed for three weeks, once a week, on the same day and time of the week.
  Fatigue index was calculated by the following equation: FI(%)= (STmean / STbest x 100) ˗ 100 to measure the percentage of decrease in performance between all sprints. One of the variables from BST to evaluate performance.

SECONDARY OUTCOMES:
Questionnaire of fatigue | This questionnaire was answered for the participants in the last day of the tests, so, at the end of the third week of the tests.
  A quick perception of fatigue survey. The questionnaire consisted of eight questions pertaining to perception of training, sleep, leg pain, concentration, effectiveness, anxiety, irritability and stress. Each question was evaluated according to a score scale where 1-2 points corresponds to "not at all", 3-4 points to "normal", and 5-7 to "very much". The scores was calculated according to the relative importance of each question and a lower score indicates better general well-being perception, and a higher score demonstrates greater fatigue perception.
Blood Lactate analysis | Blood sample was collected in the three phases of the study (three weeks, once a week) at 3, 10, 30 and 60 minutes after BST.
  Blood samples were collected from the athlete's fingertips prior to stretching and warming-up (baseline), and at 3, 10, 30 and 60 minutes after BST at each of the three study stages/phase (exercise tests).

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar P Leal-Junior, PhD, PT, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all data is properly stored in electronic devices and available for possible doubts regarding to methodological procedures or results.

REFERENCES:
- [Result] Antonialli FC, De Marchi T, Tomazoni SS, Vanin AA, dos Santos Grandinetti V, de Paiva PR, Pinto HD, Miranda EF, de Tarso Camillo de Carvalho P, Leal-Junior EC. Phototherapy in skeletal muscle performance and recovery after exercise: effect of combination of super-pulsed laser and light-emitting diodes. Lasers Med Sci. 2014 Nov;29(6):1967-76. doi: 10.1007/s10103-014-1611-7. Epub 2014 Jun 19. PMID 24942380
- [Result] Albuquerque-Pontes GM, Vieira RP, Tomazoni SS, Caires CO, Nemeth V, Vanin AA, Santos LA, Pinto HD, Marcos RL, Bjordal JM, de Carvalho Pde T, Leal-Junior EC. Effect of pre-irradiation with different doses, wavelengths, and application intervals of low-level laser therapy on cytochrome c oxidase activity in intact skeletal muscle of rats. Lasers Med Sci. 2015 Jan;30(1):59-66. doi: 10.1007/s10103-014-1616-2. Epub 2014 Jun 24. PMID 24957189
- [Result] Wragg CB, Maxwell NS, Doust JH. Evaluation of the reliability and validity of a soccer-specific field test of repeated sprint ability. Eur J Appl Physiol. 2000 Sep;83(1):77-83. doi: 10.1007/s004210000246. PMID 11072777
- [Result] Johnston RD, Gabbett TJ, Jenkins DG. Applied sport science of rugby league. Sports Med. 2014 Aug;44(8):1087-100. doi: 10.1007/s40279-014-0190-x. PMID 24748460